CLINICAL TRIAL: NCT07232030
Title: Barostim-Enabled NEurohormonal Intervention For Improving Treatment of Heart Failure (BENEFIT-HF)
Brief Title: Barostim-Enabled NEurohormonal Intervention For Improving Treatment of Heart Failure
Acronym: BENEFIT-HF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CVRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 360069-001
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure; Heart Failure NYHA Class II; Heart Failure NYHA Class III
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled, multicenter clinical trial. Eligible participants will be randomized in a 2:1 ratio to receive Baroreflex Activation Therapy (BAT) with an implanted Barostim System in addition to usual care medical management (Device Arm) or to receive usual care medical management alone with no device implant (Control Arm).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Device Arm (Experimental): Participants will receive Baroreflex Activation Therapy (BAT) with an implanted Barostim System in addition to usual care medical management.
  Interventions: Device: Barostim System
- Control Arm (Active Comparator): Participants will receive usual care medical management alone with no Barostim System device implant.
  Interventions: Other: Usual care medical management

INTERVENTIONS:
Device: Barostim System — Baroreflex Activation Therapy (BAT) using the Barostim System
  Arms: Device Arm
Other: Usual care medical management — Usual care medical management alone - no device implant
  Arms: Control Arm

SUMMARY:
The purpose of BENEFIT-HF is to demonstrate the safety and effectiveness of Baroreflex Activation Therapy (BAT) with the Barostim System in participants with heart failure, defined as NYHA Functional Class II or III, LVEF < 50% and NT-proBNP < 5,000 pg/mL despite being treated with Guideline-Directed Medical Therapies (medications and devices). It includes demonstration that treatment with the Barostim System, relative to usual care medical management, reduces the rate of all-cause mortality and Heart Failure Morbidity (Cardiac Transplant, Durable LVAD, or Worsening Heart Failure Events).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or above
2. NYHA Functional Class II or III heart failure symptoms at the time of screening
3. Left ventricular ejection fraction < 50% within 6 months of consent
4. Heart failure accompanied by either:

   * Screening local lab NT-proBNP ≥ 400 AND < 5,000 pg/mL or a BNP ≥100 AND < 1,250 pg/mL, adjusted for BMI in a stable outpatient setting OR
   * A documented Worsening Heart Failure Event in the 6 months prior to or concurrent with consent, AND an NT-proBNP < 5,000 pg/mL or BNP < 1,250 pg/mL, adjusted for BMI in a stable outpatient setting.

   Note: If participant is taking sacubitril/valsartan (i.e. Entresto®), NT-proBNP must be used for screening eligibility. NT-proBNP and BNP to be adjusted for BMI using a 4% reduction per BMI unit over 25 kg/m2.
5. On optimal, maximally tolerated Guideline Directed Medical Therapy (GDMT) (medications and devices) per current country specific guidelines (e.g. US follows AHA/ACC guidelines, Germany follows DGK/ESC guidelines) for the treatment of heart failure, when appropriate, throughout screening/baseline evaluation and for at least 4 weeks prior to consent:

   * No more than a 100% increase or a 50% decrease of the dosage of any one medication other than an oral diuretic.
   * Medication changes within a drug class are allowed as long as the equivalent dosage is within the limits specified above.
   * Unrestricted changes in oral diuretics are allowed.
   * For participants with LVEF between 40-50%, SGLT2 inhibitors and mineralocorticoid receptor antagonists (MRAs) are encouraged and should be initiated before consent when possible.
6. Six-minute hall walk (6MHW) ≥ 100 m AND ≤ 450 m within 15 days prior to randomization.
7. If female and of childbearing potential, must have a negative pregnancy test within 15 days prior to randomization.
8. Be an appropriate candidate for the trial and the surgical procedure as determined by the investigator or designee and the surgeon.
9. Have signed an informed consent form for participation in this trial.

Exclusion Criteria:

1. Any contraindications to Barostim as noted in Instructions for Use.
2. An existing device which contraindicates Barostim specifically or unipolar therapy in general.
3. Advanced heart failure defined by any of the following:

   * AHA/ACC Stage D heart failure.
   * Two or more NT-proBNP results >5,000 pg/mL or BNP >1,250 pg/mL in a stable outpatient setting within 3 months prior to consent. If participant is taking sacubitril/valsartan (i.e. Entresto®), NT-proBNP must be used for screening eligibility.
   * Current or prior continuous or intermittent intravenous positive inotrope therapy.
   * Has received, is receiving, or scheduled to receive LVAD therapy.
   * Solid organ or hematologic transplant or currently being evaluated for cardiac transplant.
4. Serum estimated glomerular filtration rate (eGFR) < 20 mL/min/1.73 m2 or has end-stage renal disease.
5. Recurring symptomatic hypotension.
6. Life expectancy less than one year.
7. An inappropriate trial candidate as evidenced by at least one of the following:

   * Has received or is receiving chronic dialysis.
   * Is within WHO groups 1, 3, 4, or 5 pulmonary hypertension.
   * Severe COPD or severe restrictive lung disease requiring chronic oral steroid use or any oxygen use.
   * Heart failure secondary to a reversible cause, such as cardiac structural valvular disease, acute myocarditis and pericardial constriction.
   * Active malignancy with the exception of non-melanoma skin cancers.
   * Infiltrative cardiomyopathy (e.g. cardiac amyloidosis).
   * Any other serious medical condition that may adversely affect the safety of the participant or validity of the trial, in the opinion of the investigator.
8. Any of the following within 3 months prior to consent:

   * Myocardial infarction
   * Unstable angina
   * Percutaneous coronary intervention (e.g. PTCA)
   * Cerebral vascular accident or transient ischemic attack
   * Cardiac arrest
   * Surgical cardiac intervention (e.g., CABG, cardiac ablation, valve replacement, CRT/ICD implantation, IPG battery replacements)
9. Surgery planned to occur within 45 days of the Barostim implant procedure. This includes pacemaker or ICD implants or battery replacements.
10. Enrolled and active in another clinical trial (e.g. device, pharmaceutical, or biological) unless approved by the CVRx Clinical Research department.
11. Unable or unwilling to fulfill the Protocol medication compliance and follow-up requirements, for reasons including but not limited to an unresolved history of alcohol or substance abuse or psychiatric disorder. Participant is a member of a vulnerable population who, in the judgment of the investigator, is unable to give Informed Consent for reasons of incapacity, immaturity, adverse personal circumstances or lack of autonomy. This may include individuals with mental disability, persons in nursing homes, impoverished persons, persons in emergency situations, homeless persons, nomads, refugees, and those permanently incapable of giving informed consent. Vulnerable populations also include university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces, and persons kept in detention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2033-01 (Estimated); Study Completion 2033-01 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint | Through 24-months follow-up
  Composite of all-cause mortality and Heart Failure Morbidity, defined as Cardiac Transplant, Durable LVAD, or Worsening Heart Failure Events, assessed through 24 months of follow-up.
Primary Safety Endpoint | Within 180 days of the device implant
  The event-free rate of all system- and procedure-related Major Adverse Neurological and Cardiovascular Events (MANCE) occurring within 180 days of the device implant, assessed among participants who were randomized to the Device Arm and in whom an implant has been achieved or attempted.

SECONDARY OUTCOMES:
Quality of Life (QoL) Score Change | 12-months follow-up
  QoL score change, as measured by the Minnesota Living With Heart Failure (MLWHF) questionnaire from baseline to 12 months.
6MHW distance change | 12-months follow-up
  6-minute hall walk (6MHW) distance change from baseline to 12 months.
Days lost to death or hospitalization | 24-months follow-up
NT-proBNP level change | 12-months follow up
  NT-proBNP level change from baseline to 12 months
All-cause mortality | 24-months follow-up

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor website — https://www.cvrx.com/